CLINICAL TRIAL: NCT04647058
Title: Randomized Controlled Trial of Supercharged End-to-Side (SETS) Anterior Interosseous Nerve Transfer for Severe Cubital Tunnel Syndrome
Brief Title: Randomized Trial of Supercharged End-to-Side Anterior Interosseous Nerve Transfer for Severe Cubital Tunnel Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Philip Blazar (Unknown); Matthew J. Carty (Unknown); Arriyan S. Dowlatshahi (Unknown); George S. M. Dyer (Unknown); Brandon E. Earp (Unknown); Carl M. Harper (Unknown); Lydia A. Helliwell (Unknown); Tamara D. Rozental (Unknown); Christian E. Sampson (Unknown); Simon G. Talbot (Unknown)
Responsible Party: Principal Investigator, Dafang Zhang, M.D., Instructor in Orthopaedic Surgery, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020P003713
Record Dates: First submitted 2020-11-16; First posted 2020-11-30 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Cubital Tunnel Syndrome; Ulnar Nerve Compression; Ulnar Nerve Palsy; Ulnar Nerve Entrapment; Ulnar Nerve Entrapment at Elbow; Ulnar Nerve Entrapment Syndrome; Ulnar Neuropathies; Ulnar Claw
Keywords: cubital tunnel syndrome; ulnar nerve compression; cubital tunnel release; cubital tunnel decompression; supercharged end-to-side; SETS; anterior interosseous nerve transfer
MeSH Terms: conditions — Cubital Tunnel Syndrome; Ulnar Nerve Compression Syndromes; Ulnar Neuropathies | interventions — Nerve Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cubital tunnel release (Active Comparator): The control group will undergo cubital tunnel release in situ. In cases of preoperative or intraoperative ulnar nerve instability, anterior transposition of the ulnar nerve will be performed.
  Interventions: Procedure: Cubital tunnel release
- Supercharged end-to-side (SETS) nerve transfer (Experimental): The SETS group will undergo the same procedure as described above, with the addition of the SETS procedure consisting of a end-to-side transfer of the anterior interosseous nerve to the ulnar nerve motor branch. Decompression of Guyon's canal during the SETS procedure is at the discretion of the treating surgeon.
  Interventions: Procedure: Supercharged end-to-side (SETS) nerve transfer

INTERVENTIONS:
Procedure: Cubital tunnel release — The control group will undergo cubital tunnel release in situ. In cases of preoperative or intraoperative ulnar nerve instability, anterior transposition of the ulnar nerve will be performed.
  Arms: Cubital tunnel release
Procedure: Supercharged end-to-side (SETS) nerve transfer — The SETS group will undergo the same procedure as described above, with the addition of the SETS procedure consisting of a end-to-side transfer of the anterior interosseous nerve to the ulnar nerve motor branch. Decompression of Guyon's canal during the SETS procedure is at the discretion of the treating surgeon.
  Arms: Supercharged end-to-side (SETS) nerve transfer

SUMMARY:
Functional motor recovery distal to a peripheral nerve lesion is predicated upon time to reinnervation of the motor end plate and the number of regenerate axons that reach the target. Supercharged end-to-side (SETS) transfer of the anterior interosseous nerve to the motor fascicle of the ulnar nerve at the level of the distal forearm has been proposed as an adjunct procedure in severe cubital tunnel syndrome to augment motor recovery of the ulnar-innervated intrinsic muscles. Multiple Level IV Therapeutic studies and a systematic review of Level IV Therapeutic studies have reported favorable clinical and electrodiagnostic outcomes following SETS for cubital tunnel syndrome, with low rates of complications. However, in the absence of controls, it remains unclear what proportion of the observed intrinsic motor recovery is attributable to the SETS procedure. The objective of this randomized trial is to compare the results of ulnar nerve decompression with or without SETS for severe cubital tunnel syndrome.

DETAILED DESCRIPTION:
Null hypothesis: Ulnar nerve decompression with or without supercharged end-to-side (SETS) anterior interosseous nerve transfer for McGowan classification stage III cubital tunnel syndrome results in similar ulnar intrinsic motor recovery.

Background Functional motor recovery distal to a peripheral nerve lesion is predicated upon time to reinnervation of the motor end plate and the number of regenerate axons that reach the target. Supercharged end-to-side (SETS) transfer of the anterior interosseous nerve to the motor fascicle of the ulnar nerve at the level of the distal forearm has been proposed as an adjunct procedure in severe cubital tunnel syndrome to augment motor recovery of the ulnar-innervated intrinsic muscles. The proposed mechanism of action of SETS is twofold: (1) "babysitting" the motor end plates until native regenerate axons reach their target, and (2) augmented partial recovery through axonal growth through the new pathway.

Multiple Level IV Therapeutic studies and a systematic review of Level IV Therapeutic studies have reported favorable clinical and electrodiagnostic outcomes following SETS for cubital tunnel syndrome, with low rates of complications. However, in the absence of controls, it remains unclear what proportion of the observed intrinsic motor recovery is attributable to the SETS procedure. Koriem et al. recently published a prospective, randomized comparative study of ulnar nerve repair with or without SETS for proximal ulnar nerve injuries and demonstrated superior intrinsic recovery and claw correction with the SETS procedure. Prospective, randomized trials of SETS for severe cubital tunnel syndrome are needed.

The objective of this study is to compare the results of ulnar nerve decompression with or without SETS for severe cubital tunnel syndrome. In this study, severe cubital tunnel syndrome is defined as McGowan classification stage III disease (sensory deficits, motor deficits, and the presence of intrinsic atrophy).

Methods Patient Selection A prospective, randomized controlled trial will be conducted at two participating institutions: Brigham and Women's Hospital and Beth Israel Deaconess Medical Center. Inclusion criteria are patients 18 years of age or older indicated for surgical treatment of severe cubital tunnel syndrome at one of the two participating institutions. Inclusion criteria furthermore includes a preoperative nerve conduction study and electromyography documenting ulnar neuropathy at the elbow with present fibrillations and positive sharp waves in the FDI or ADM within one year of surgery. Severe cubital tunnel syndrome is defined in this study as McGowan classification stage IIB or III disease (sensory deficits, motor deficits, and the presence of intrinsic atrophy). Exclusion criteria include ulnar nerve transections, traumatic brachial plexus injuries, brachial plexus neuritis (e.g. Parsonage-Turner), cervical radiculopathy, primary motor neuropathy (e.g. Charcot-Marie-Tooth), prior cubital tunnel surgery, and oncologic etiologies of ulnar nerve compression. Exclusion criteria additionally include patients who are not capable of decision-making or are unable to understand the study procedures. Non-English speaking patients are excluded since our secondary outcome variables may not have been translated and validated in other language(s). Comorbid carpal tunnel syndrome, concomitant carpal tunnel release, comorbid diabetes mellitus, and internervous connections such as Martin-Gruber connections are not criteria for exclusion.

Randomization Patients included in this study will be randomly assigned to the SETS group or the control group with a 1:1 enrollment ratio. A computerized random number generator will be used for allocation, which will be concealed by sequentially numbered, sealed, opaque envelopes opened after patient consent and enrollment.

Treatment The control group will undergo cubital tunnel release in situ. In cases of preoperative or intraoperative ulnar nerve instability, anterior transposition of the ulnar nerve will be performed. A soft dressing will be applied for in situ decompressions. A posterior elbow plaster splint will be used for anterior transpositions for 2 weeks. Patients will receive formal occupational therapy for scar massage, range of motion, and progressive intrinsic strengthening starting at 2 weeks postoperatively for 6 weeks duration.

The SETS group will undergo the same procedure as described above, with the addition of the SETS procedure as previously described.1 Decompression of Guyon's canal during the SETS procedure is at the discretion of the treating surgeon. In addition to the aforementioned elbow dressing, a neutral wrist splint will be used for 2 weeks. Patients will receive formal occupational therapy for scar massage, range of motion, and motor re-education consisting of repetitive forearm pronation exercises starting at 2 weeks postoperatively for 6 weeks duration.

Data collection

Primary outcome variable:

Subterminal key pinch strength (kg) - continuous Time points: 0, 3 months, 6 months, 12 months, 18 months

Secondary outcome variables:

Patient-Rated Ulnar Nerve Evaluation (PRUNE) score - continuous, non-parametric Disabilities of the Arm, Shoulder and Hand (DASH) score - continuous, non-parametric MRC forearm pronation strength in elbow flexion and extension - ordinal, non-parametric Time points: 0, 3 months, 6 months, 12 months, 18 months

Explanatory variables:

Age - continuous, non-parametric Sex - dichotomous Dominant hand - dichotomous BMI - continuous, parametric Diabetes mellitus - dichotomous Smoking status - dichotomous Worker's Compensation status - dichotomous Duration of symptoms at presentation (months) - continuous, non-parametric Preoperative NCS SNAP - continuous, parametric Preoperative NCS CMAP - continuous, parametric Guyon's canal decompression - dichotomous

Statistical analysis An a priori power calculation was performed. Assuming a 1:1 enrollment ratio and a mean subterminal key pinch strength of 4 kg (standard deviation 1 kg), a sample size of 32 (16 patients in each group) has 80% power to detect a 1 kg difference in subterminal key pinch strength between groups.

Descriptive statistics will be calculated for the study cohorts. The student's t-test will be used to compare the primary outcome variable and the Mann-Whitney U test will be used to compare the secondary outcome variables between the SETS group and the control group.

The investigators will use bivariate analysis to screen for factors associated with poorer outcome in the SETS group and in the control group. Variables that meet our inclusion criteria (p < 0.1) will be included in a multiple regression model to assess for independent factors associated with poorer outcomes following the study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Severe cubital tunnel syndrome is defined in this study as McGowan classification stage IIB or III disease (sensory deficits, motor deficits, and the presence of intrinsic atrophy)
* Indicated for surgical treatment of severe cubital tunnel syndrome at one of the two participating institutions
* Preoperative nerve conduction study and electromyography documenting ulnar neuropathy at the elbow with present fibrillations and positive sharp waves in the FDI or ADM within one year of surgery

Exclusion Criteria:

* Ulnar nerve transections
* Traumatic brachial plexus injuries
* Brachial plexus neuritis (e.g. Parsonage-Turner)
* Cervical radiculopathy
* Primary motor neuropathy (e.g. Charcot-Marie-Tooth)
* Prior cubital tunnel surgery
* Oncologic etiologies of ulnar nerve compression
* Patients who are not capable of decision-making or are unable to understand the study procedures
* Non-English speaking patients are excluded since our secondary outcome variables may not have been translated and validated in other language(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Subterminal key pinch strength | 18 months
  The primary outcome variable of this study is subterminal key pinch strength assessed by dynanometer measured in kg. Subterminal key pinch strength is a direct assessment of ulnar-innervated muscle strength.

SECONDARY OUTCOMES:
Patient-Rated Ulnar Nerve Evaluation (PRUNE) score | 18 months
  The PRUNE score is a validated patient-reported outcome measure of ulnar nerve function. The total PRUNE score ranges from 0 to 100, with 0 denoting no symptoms and 100 denoting the worst possible symptoms.
Disabilities of the Arm, Shoulder and Hand (DASH) score | 18 months
  The DASH score is a validated patient-reported outcome measure of upper extremity function. The total DASH score ranges from 0 to 100, with 0 denoting no disability and 100 denoting the most severe disability.
MRC forearm pronation strength | 18 months
  The MRC forearm pronation strength is a commonly used physician-rated scoring system for muscle strength on a 0 to 5 scale and will be used to assess donor deficits from an anterior interosseous nerve transfer, with 0 denoting no strength and 5 denoting full strength.

CONTACTS AND LOCATIONS:
Overall Officials: Dafang Zhang, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour J, Yee A, Kahn LC, Mackinnon SE. Supercharged end-to-side anterior interosseous to ulnar motor nerve transfer for intrinsic musculature reinnervation. J Hand Surg Am. 2012 Oct;37(10):2150-9. doi: 10.1016/j.jhsa.2012.07.022. PMID 23021177
- [Background] Jarvie G, Hupin-Debeurme M, Glaris Z, Daneshvar P. Supercharge End-to-Side Anterior Interosseous Nerve to Ulnar Motor Nerve Transfer for Severe Ulnar Neuropathy: Two Cases Suggesting Recovery Secondary to Nerve Transfer. J Orthop Case Rep. 2018 Sep-Oct;8(5):25-28. doi: 10.13107/jocr.2250-0685.1194. PMID 30740369
- [Background] Davidge KM, Yee A, Moore AM, Mackinnon SE. The Supercharge End-to-Side Anterior Interosseous-to-Ulnar Motor Nerve Transfer for Restoring Intrinsic Function: Clinical Experience. Plast Reconstr Surg. 2015 Sep;136(3):344e-352e. doi: 10.1097/PRS.0000000000001514. PMID 26313839
- [Background] Dengler J, Dolen U, Patterson JMM, Davidge KM, Kahn LC, Yee A, Mackinnon SE. Supercharge End-to-Side Anterior Interosseous-to-Ulnar Motor Nerve Transfer Restores Intrinsic Function in Cubital Tunnel Syndrome. Plast Reconstr Surg. 2020 Oct;146(4):808-818. doi: 10.1097/PRS.0000000000007167. PMID 32590517
- [Background] Dunn JC, Gonzalez GA, Fernandez I, Orr JD, Polfer EM, Nesti LJ. Supercharge End-to-Side Nerve Transfer: Systematic Review. Hand (N Y). 2021 Mar;16(2):151-156. doi: 10.1177/1558944719836213. Epub 2019 Mar 29. PMID 30924361
- [Background] Koriem E, El-Mahy MM, Atiyya AN, Diab RA. Comparison Between Supercharged Ulnar Nerve Repair by Anterior Interosseous Nerve Transfer and Isolated Ulnar Nerve Repair in Proximal Ulnar Nerve Injuries. J Hand Surg Am. 2020 Feb;45(2):104-110. doi: 10.1016/j.jhsa.2019.11.005. Epub 2019 Dec 20. PMID 31866151
- [Background] MacDermid JC, Grewal R. Development and validation of the patient-rated ulnar nerve evaluation. BMC Musculoskelet Disord. 2013 Apr 26;14:146. doi: 10.1186/1471-2474-14-146. PMID 23617407
- [Background] Bertelli JA. Subterminal key pinch dynamometry: a new method to quantify strength deficit in ulnar nerve paralysis. J Hand Surg Eur Vol. 2020 Oct;45(8):813-817. doi: 10.1177/1753193420919283. Epub 2020 Apr 29. PMID 32349609
- [Background] Head LK, Zhang ZZ, Hicks K, Wolff G, Boyd KU. Evaluation of Intrinsic Hand Musculature Reinnervation following Supercharge End-to-Side Anterior Interosseous-to-Ulnar Motor Nerve Transfer. Plast Reconstr Surg. 2020 Jul;146(1):128-132. doi: 10.1097/PRS.0000000000006903. PMID 32590654